CLINICAL TRIAL: NCT03361150
Title: High-Intensity Interval Training Versus Moderate Continuous Training in Multimodal Prehabilitation for Colorectal Surgery: A Randomized Controlled Trial.
Brief Title: High-Intensity Interval vs. Moderate Continuous Training in Surgical Prehabilitation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Franco Carli, Clinical Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-244-MUHC
Record Dates: First submitted 2017-11-23; First posted 2017-12-04 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Cancer; Physical Activity
Keywords: prehabilitation
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIT (Experimental): Preoperative nutrition, relaxation strategies + high intensity interval training (HIT). HIT alternates a series of high-intensity bouts with relief period. This will be a personalized, 3 times per week, 40-min exercise. Protein supplement will be prescribed if needed to achieve a daily intake of 1.5 g protein/kg.
  Interventions: Procedure: HIT
- MCT (Active Comparator): Preoperative nutrition, relaxation strategies + high intensity interval training (MCT). MCT is continuous exercise with a constant intensity below anaerobic threshold. This will be a personalized, 3 times per week, 40-min exercise. Protein supplement will be prescribed if needed to achieve a daily intake of 1.5 g protein/kg.
  Interventions: Procedure: MCT

INTERVENTIONS:
Procedure: HIT — Both exercise protocol will be personalized, 3 times per week, 40-min exercise. HIT alternates a series of high-intensity bouts with relief period. MCT is continuous exercise with a constant intensity below anaerobic threshold.
  Arms: HIT
Procedure: MCT — Both exercise protocol will be personalized, 3 times per week, 40-min exercise. MCT is continuous exercise with a constant intensity below anaerobic threshold.
  Arms: MCT

SUMMARY:
Surgery is a stressful procedure associate with perioperative physical impairment. In a previous study, the investigators showed that physical fitness could be optimize in surgical patients using prehabilitation, a preoperative conditioning intervention in form of exercise, nutrition and relaxation technique. The best modality of exercise has yet to be known.The purpose of this study is to compare high interval (HIT) vs. moderate continuous intensity (MC) training, integrated in a prehabilitation intervention in colorectal surgical patients.

DETAILED DESCRIPTION:
All patients will receive prehabilitation preoperatively for 4 weeks, that is composed of 3 elements, exercise, nutritional supplements and psychological coping strategies. Both exercise protocol will be supervised, 3-time per week, in-hospital programs. Patients will be randomized to perform either HIT or MC training. Exercise intensity will be defined and personalized on the individual values at cardiopulmonary exercise testing (CPET). Patients' nutritional status and dietary intake will be assessed by the nutritionist, and supplement will be prescribed if needed to achieve a daily intake of 1.5 g protein/kg. Perioperative care will follow the McGill Surgical Recovery Pathway, also called Enhanced Recovery Program, which is an evidence-based care plan set up by the Surgical Recovery (SuRe) multidisciplinary committee of the McGill University Health Centre.

ELIGIBILITY:
Inclusion Criteria:

* Subjects eligible to enter the study will include those aged 18 and above and referred electively for resection of malignant colorectal lesions.

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) health status class 4-5 or co-morbid medical, physical and mental conditions interfering with the ability to perform exercise at home or to complete the testing procedures. Poor English and French comprehension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Oxygen consumption (VO2) | 4 weeks (before surgery)
  Cardiopulmonary exercise testing (CPET) will be conducted on a cycle ergometer. Coupling expired gas analysis with minute ventilation, It will provide oxygen consumption during exercise.

SECONDARY OUTCOMES:
Six-minute walking distance. | 4 weeks (before surgery)
  Using a 6-minute walk test, subjects are instructed to walk back and forth, in a 20 m stretch of hallway, for six minutes, at a pace that would make them tired by the end of the walk.
Sit-to-Stand test | 4 weeks (before surgery)
  Sit-to-Stand test is measured by the Senior Fitness Test, to assess an individuals lower-body strength. This is done by having the individual sit on a chair and attempt to stand as many times in a maximum of 30 seconds.
Community Health Activities Model Program for Seniors (CHAMPS) score | 4 weeks (before surgery)
  Physical activity level will be measured through the Community Health Activities Model Program for Seniors (CHAMPS) questionnaire. The CHAMPS is a self-reported measure of physical activity, comprising 41 activities evaluated according to the total number of hours done during an average week. Each physical activity is assigned a MET (metabolic equivalent) value yielding average weekly caloric expenditure for the listed physical activities. Continuos variable, measured in kcal/week, minimum score 3.5, higher value from baseline will represent a better outcome.
Hospital Anxiety and Depression Scale (HADS) score | 4 weeks (before surgery)
  Depression and anxiety will be assessed by the Hospital Anxiety and Depression Scale (HADS), a 14-question measure with seven items each for depression and anxiety. HADS generates separate scores for anxiety and depression as well as a combined score of psychological distress. Continuos variable 0-21 (0-7 normal value, 11-21 anxiety/depression), higher value from baseline will represent a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gillis C, Li C, Lee L, Awasthi R, Augustin B, Gamsa A, Liberman AS, Stein B, Charlebois P, Feldman LS, Carli F. Prehabilitation versus rehabilitation: a randomized control trial in patients undergoing colorectal resection for cancer. Anesthesiology. 2014 Nov;121(5):937-47. doi: 10.1097/ALN.0000000000000393. PMID 25076007
- [Derived] Minnella EM, Ferreira V, Awasthi R, Charlebois P, Stein B, Liberman AS, Scheede-Bergdahl C, Morais JA, Carli F. Effect of two different pre-operative exercise training regimens before colorectal surgery on functional capacity: A randomised controlled trial. Eur J Anaesthesiol. 2020 Nov;37(11):969-978. doi: 10.1097/EJA.0000000000001215. PMID 32976204